CLINICAL TRIAL: NCT03283514
Title: Esthetic Expectations of Edentulous Patients Followed in a French Dental Clinic
Status: Completed | Type: Observational
Sponsor: Hôpital Rothschild (Other)
Responsible Party: Principal Investigator, Dr Braud Adeline, maitre de conférences -praticien hospitalier, Hôpital Rothschild
Other Study IDs: 01
Record Dates: First submitted 2017-09-09; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Complete Edentulism
MeSH Terms: interventions — Denture, Complete

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Complete denture — questionnaire

SUMMARY:
Esthetic is a major factor in complete denture (CD) success. Patient involvement in esthetic project plays a crucial role in denture acceptance and patient satisfaction. Historically, teeth choice and arrangement were made according to Frush and Ficher's recommendations focusing on natural looking of esthetics. Dentists may also propose to restore the dentate state looking for denture when preextraction data are available. Recently, a patient-centered approach based on attractivity has been proposed and may lead to in an appearance transcending the laws of nature.

The aim of the present study was to investigate actual denture esthetic expectations in a French edentate population followed in a university dental clinic (Rothschild Hospital , AP-HP).

DETAILED DESCRIPTION:
Inclusion criteria : being currently edentulous within at least within the maxillary arch, literate French speakers, willing and able to complete the survey in a single sitting. Clinical data collection was made by a unique examiner and concerned length of edentulism, antagonist arch, existence of preextraction data, smile attractivity opinion. The respondents completed a questionnaire identifying their age, sex, educational and income level. Patients were also asked for their denture look preference among 4 esthetic projects: 1) restoring pre-extraction (dentate) looking, 2) restoring actual denture looking, 3) creating natural looking, 4) creating perfect looking, 5) no opinion. Each project was explained similarly by the same examiner. Statistical analysis using a Pearson Chi-squared test at a 0.05 level of significance was conducted for associations between esthetic projects preference and tested variables.

ELIGIBILITY:
Inclusion criteria : Currently edentulous maxillary arch, literate French speakers, willing and able to complete the survey in a single sitting. Inclusion Criteria:

Exclusion Criteria: Aged under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Totally edentulous subjects (20 women, 22 men, mena aged: 67.9 ± 12.2 years) attending maxillary CD in the department of prosthodontics of the Hopital Rothschild (AP-HP) are concerned by recruitment and are proposed to participate.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
esthetic preferred project | Esthetic expectation evaluated at date of inclusion
  Patients were asked for their denture-looking expectations among 4 esthetic projects: 1) restoring pre-extraction dentate looking, 2) restoring actual denture looking, 3) creating natural looking, 4) creating perfect looking, 5) no opinion.

SECONDARY OUTCOMES:
age | evaluated at date of inclusion
  Respondents completed a questionnaire identifying their age (in years)
gender | evaluated at date of inclusion
  Respondents completed a questionnaire identifying their gender (man or woman)
educational level | evaluated at date of inclusion
  Respondents completed a questionnaire identifying their educational level : last degree (no degree at al, French General Certificate Secondary Education, High School Diploma, Vocational Training Certificate taken at Secondary School, university degree)
month income level, | evaluated at date of inclusion
  Respondents completed a questionnaire identifying their income level each month : in euros
length of edentulism, | evaluated at date of inclusion
  Respondents completed a questionnaire identifying the duration of edentulism (in years)
smile attractivity opinion | evaluated at date of inclusion
  Respondents completed a questionnaire identifying their smile attractivity opinion Respondents completed a questionnaire identifying the most attractive smile among 4 esthetic situations : preextraction-looking smile, denture-like smile, natural-like smile, perfect smile.
preextraction data available | evaluated at date of inclusion
  Respondents completed a questionnaire identifying the existence of preextraction data available (available or not available)

IPD SHARING:
Plan to Share IPD: Undecided